CLINICAL TRIAL: NCT02867631
Title: A Randomized Controlled Trial (RCT) of an Intervention to Combat Postpartum Weight Retention
Brief Title: Postpartum Weight Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Aetna, Inc. (Industry)
Responsible Party: Principal Investigator, Charmaine Smith Wright, Principle Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 815827
Record Dates: First submitted 2015-05-29; First posted 2016-08-16 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Obesity; Hypertension; Depression
Keywords: Intervention study; Maternal obesity; Nutrition; Maternal child health
MeSH Terms: conditions — Obesity; Hypertension; Depression; Pregnancy in Obesity | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced control (No Intervention): Regular care as provided by the community based organization from which the convenience sample is recruited with one year of assessments only
- Intervention (Experimental): 6 week challenge with 1 year of home visits: health texting, in home exercise supports, social support, healthy eating and feeding classes
  Interventions: Behavioral: 6 week challenge with 1 year of home visits: health texting, in home exercise supports, social support, healthy eating and feeding classes

INTERVENTIONS:
Behavioral: 6 week challenge with 1 year of home visits: health texting, in home exercise supports, social support, healthy eating and feeding classes — 6 week challenge with 1 year of home visits: health texting, in home exercise supports, social support, healthy eating and feeding classes
  Arms: Intervention

SUMMARY:
The Postpartum Weight Management Study is a true community-academic collaboration, bringing together Maternity Care Coalition (MCC) staff and the investigator, Dr. Charmaine Smith Wright from the University of Pennsylvania to address the needs of postpartum moms. The project is an innovative intervention to help moms lose weight after the birth of their baby. Helping mothers control their weight during pregnancy and beyond can help both mother and baby avoid later obesity and cardiovascular disease. Although all women are at risk for retaining the weight gained during pregnancy, this problem is amplified for low-income, minority women. The holistic approach aims to prevent postpartum weight retention and increase breastfeeding duration with a multi-component, low-cost intervention that provides: 1) Motivational appeals delivered in text message format; 2) Environmental aides, such as a baby carrier to combine exercise with infant care, and a pedometer to accurately measure exercise at home; 3) Enhanced peer support, including home visits and group classes with other mothers; and 4) Task-oriented professional support from nutrition and lactation experts, who assist women in developing a personalized health plan. The effectiveness of the intervention will be evaluated using a randomized control methodology among clients of MCC.

ELIGIBILITY:
Inclusion Criteria:

* All women who speak English, and are within six weeks of delivering a live, term, single infants

Exclusion Criteria:

* Women who have multiple births or preterm (<38 weeks gestation) infants

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postpartum weight change | Baseline and 1 year post intervention
  Weight difference at one year post intervention and start of intervention

SECONDARY OUTCOMES:
Postpartum weight change | Baseline and 6 months post intervention start
  Weight difference at 6 months post intervention and start of intervention
Depression | Baseline, 6 weeks, 6 months, and 1 year post intervention start
  Using Edinburgh perinatal depression screen score, as a continuous and dichotomous (Yes/No) variable
Dietary quality | Baseline, 6 weeks, 6 months, and 1 year post intervention
  Descriptive analysis of a food log from the time points proposed
Infant growth | Baseline, 6 weeks, 6 months, and 1 year post intervention start
  Infant weight for length percentile at 6 weeks, 6 months, and 1 year post intervention (weight in pounds and length in inches converted to weight for length percentile using World Health Organization software support http://www.who.int/childgrowth/software/readme_stata.pdf?ua=1)
Nutrition knowledge score change | Baseline, 6 weeks, 6 months, and 1 year post intervention start
  Using validated nutrition knowledge scale at 6 weeks, 6 months, and 1 year post intervention, difference from baseline
Waist circumference as continuous measure, in inches | Baseline, 6 weeks, 6 months, and 1 year post intervention start
  Acquired at study assessments at the proposed time points
Back to prepregnancy weight | baseline and 1 year post intervention
  Dichotomous (yes/no) variable describing whether the subject returned to pre-pregnancy weight (difference between 1 year post and self-reported pre-pregnancy weight at baseline time point survey=0) or not
Back to pregnancy weight, continuous | baseline and 1 year postpartum
  Continuous (difference in 1 year post-intervention weight and self-reported pre-pregnancy weight reported at baseline time point survey) variable describing the change in weight over time

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Wright, MD MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- Maternity Care Coalition, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wright C, Mogul M, Acevedo G, Aysola J, Momplaisir F, Schwartz S, Shea J. Preparing for a trial to test a postpartum weight retention intervention among low income women: feasibility of a protocol in a community-based organization. BMC Womens Health. 2018 Jan 25;18(1):27. doi: 10.1186/s12905-018-0517-0. PMID 29370795